CLINICAL TRIAL: NCT01670188
Title: Sequential Pneumatic Compression to Prevent PICC-related Upper Extremity Venous Thrombosis in Critically Ill Neurological Patients
Brief Title: SCD Use to Prevent Deep Venous Thrombosis (DVT) in Patients With PICC Lines
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis: patients treated with SCD had higher incidence of DVT.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Alejandro Rabinstein, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12-004676
Record Dates: First submitted 2012-08-16; First posted 2012-08-22 (Estimated); Results first posted 2018-01-09 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2017-08

CONDITIONS: Deep Vein Thrombosis
Keywords: Pneumatic sequential compression device (SCD); Peripherally Inserted Central Catheters (PICC)
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Pneumatic SCD (Active Comparator): Use of pneumatic SCD (VenaFlow System - DJO Global) on upper extremity with PICC line inserted.
  Interventions: Device: Pneumatic SCD - VenaFlow System (DJO Global)
- Non-SCD group (No Intervention): Standard care

INTERVENTIONS:
Device: Pneumatic SCD - VenaFlow System (DJO Global)
  Other Names: VenaFlow System (DJO Global)
  Arms: Pneumatic SCD

SUMMARY:
The purpose of this study is to see if a compression device on the arm where a peripherally inserted central catheter (PICC) line has been inserted can prevent the formation of a blood clot around the PICC line.

DETAILED DESCRIPTION:
In a pilot prospective randomized controlled trial, consecutive patients requiring placement of a PICC line in the Neuroscience intensive care unit were randomly assigned to either the SCD (intervention) group or a non SCD (control) group.

Standardized vascular access patency protocols was used in all enrolled patients. All patients had an indwelling 5 French, double lumen PICC unless additional venous access was required by the primary service. Patients randomized to the intervention arm had an SCD placed in the arm with the PICC within 24 hours of PICC placement.

Five to seven days after placement of the PICC, the patients were examined with venous duplex ultrasound of the upper extremity to assess for the presence of venous thrombosis. The patients also had the ultrasound again 12-14 days post insertion if the PICC was kept for more than 10 days. If the PICC line was removed before 5-7 days, an upper extremity ultrasound was obtained upon PICC removal. In case of suspected symptomatic venous thromboembolism, the investigations were performed according to current practice standards. Data collection was be considered complete upon removal of the PICC line.

ELIGIBILITY:
Inclusion Criteria:

* Subject's age is greater than or equal to 18 years
* Subject is patient in neuro intensive care unit at time of PICC placement

Exclusion Criteria:

* Acute trauma to the upper extremity harboring the PICC
* Current use of prophylactic anticoagulation
* Inability to fit the SCD on the arm because of arm size
* Documented previous upper extremity DVT in the arm harboring the PICC line

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2016-10-13 (Actual); Study Completion 2016-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Rabinstein, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Rabinstein AA, Hellickson JD, Macedo TA, Lewis BD, Mandrekar J, McBane RD 2nd. Sequential Pneumatic Compression in the Arm in Neurocritical Patients with a Peripherally Inserted Central Venous Catheter: A Randomized Trial. Neurocrit Care. 2020 Feb;32(1):187-192. doi: 10.1007/s12028-019-00765-w. PMID 31236782

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients requiring placement of a peripherally inserted central catheter (PICC) line in the neuroscience intensive care unit were recruited at Mayo Clinic in Rochester, Minnesota.
Pre-assignment Details: One patient randomized to the non-SCD arm died before the first ultrasound could be obtained and therefore could not be entered into the analysis.
Groups:
- Pneumatic SCD: Use of pneumatic sequential compression device (SCD) (VenaFlow System - DJO Global) on upper extremity with peripherally inserted central catheter (PICC) line inserted.
- Non-SCD Group: Patients enrolled in this group received standard care.
Period: Overall Study
Arm/Group | Pneumatic SCD | Non-SCD Group
Started | 38 | 40
Completed | 38 | 39
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pneumatic SCD | Non-SCD Group | Total
Number analyzed (Participants) | 38 | 39 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 29 | 56
  >=65 years | 11 | 10 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 26 | 49
  Male | 15 | 13 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 38 | 39 | 77

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Experienced an Ultrasonographically-confirmed Venous Thrombosis
Description: Ultrasonographically-confirmed upper extremity venous thrombosis (symptomatic and asymptomatic) in arm with PICC catheter
Time Frame: baseline to 14 days post insertion of PICC line
Measure: Count of Participants; unit: Participants
Arm/Group | Pneumatic SCD | Non-SCD Group
Number analyzed (Participants) | 38 | 39
Participants | 13 | 5
Statistical Analysis 1: Comparison: Pneumatic SCD vs Non-SCD Group; Test type: Superiority; p = 0.02, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Pneumatic SCD | Non-SCD Group
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/39
Other Adverse Events (participants affected / at risk) | 0/38 | 0/39

LIMITATIONS AND CAVEATS:
The study was terminated early because the pre-determined interim analysis showed patients treated with the SCD had higher incidence of DVT by ultrasound.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes